CLINICAL TRIAL: NCT00750373
Title: A Randomized Comparison of Early Surgery Versus Conventional Treatment Strategy in Patients With High Embolic Risk of Infective Endocarditis
Brief Title: Early Surgery Versus Conventional Treatment in Infective Endocarditis
Acronym: EASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0257
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Endocarditis
Keywords: Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional (No Intervention): Conventional Treatment based on current guidelines
- Surgery (Active Comparator): Early surgery within 48 hours of randomization
  Interventions: Procedure: Valve surgery with removal of vegetations

INTERVENTIONS:
Procedure: Valve surgery with removal of vegetations — Early valve repair or replacement with removal of vegetations within 48 hours of randomization
  Other Names: early surgery
  Arms: Surgery

SUMMARY:
There have been no prospective clinical studies in infective endocarditis comparing early surgery with the conventional treatment strategy based on current guidelines. The purpose of this prospective randomized trial is to compare clinical outcomes of early surgery versus conventional treatment strategy in patients with high embolic risk of infective endocarditis.

DETAILED DESCRIPTION:
Infective Endocarditis is still associated with high mortality (16-25%) and high incidence of embolic events (10-49%), and the optimal therapeutic strategy remains unclear. The benefit of surgery was particularly high in patients with abscess formation, periannular complications, and moderate to severe heart failure related to acute mitral or aortic regurgitation. Retrospective studies reported that valve surgery was associated with improved survival, but the benefit of early surgery has not been adequately studied due to inherent treatment biases and significant differences in baseline characteristics. Embolic indications for surgery are more controversial, and surgery is usually performed in cases of recurrent emboli and persist vegetations despite appropriate antibiotic treatment. The combined risk of early surgery and valve prosthesis needs to be balanced against the potential benefit of preventing embolism and improving survival. Risk-benefit balance changes recently to favor early surgery in patients with high embolic risk of endocarditis for the following reasons. Identification of patients with high risk of embolism becomes possible with the use of transesophageal echocardiography. Patients with vegetation length > 10 mm on transesophageal echocardiography have a significantly higher risk of embolization. With advances in surgical technique, urgent surgery is feasible with low operative mortality, and the success rate of valve repair has been increased.

To the best of our knowledge, there have been no prospective outcome studies comparing early surgery with the conventional treatment strategy based on current guidelines. The purpose of this multi-center, prospective, randomized trial is to compare clinical outcomes of early surgery versus conventional treatment strategy in patients with high embolic risks of infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as infective endocarditis based on modified Duke criteria fulfilling both conditions:

  * severe mitral or aortic regurgitation
  * vegetation length > 10 mm on mitral or aortic valve

Exclusion Criteria:

* Patients with urgent and emergent indication of surgery based on current guidelines; aortic abscess, moderate to severe heart failure due to valvular regurgitation, periannular complications, fungal endocarditis
* Prosthetic valve endocarditis
* Patient without vegetations on echocardiography
* Patients with ischemic or hemorrhagic stroke within 2 weeks before the admission
* Patients referred from other hospitals more than 7 days after the appropriate antibiotic treatment of infective endocarditis
* Patients who were not candidates for surgery based on age > 80 years and coexisting malignancies
* Patients who did not consent to participate

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-09; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Kang DH, Lee S, Kim YJ, Kim SH, Kim DH, Yun SC, Song JM, Chung CH, Song JK, Lee JW. Long-Term Results of Early Surgery versus Conventional Treatment for Infective Endocarditis Trial. Korean Circ J. 2016 Nov;46(6):846-850. doi: 10.4070/kcj.2016.46.6.846. Epub 2016 Oct 20. PMID 27826345
- [Derived] Kang DH, Kim YJ, Kim SH, Sun BJ, Kim DH, Yun SC, Song JM, Choo SJ, Chung CH, Song JK, Lee JW, Sohn DW. Early surgery versus conventional treatment for infective endocarditis. N Engl J Med. 2012 Jun 28;366(26):2466-73. doi: 10.1056/NEJMoa1112843. PMID 22738096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were eligible for enrollment if they were diagnosed as definite infective endocarditis and had both severe mitral or aortic valve disease and vegetation length > 10 mm. Between September 2006 and March 2011, a total of 76 patients were enrolled at the Asan Medical Center (n=71) and Seoul National University Hospital (n=5) in Korea.
Pre-assignment Details: The exclusion criteria were defined as patients with moderate to severe CHF; heart block; annular or aortic abscess; fungal endocarditis; and those who were not candidates for early surgery on the basis of age > 80 years, coexisting major embolic stroke with a risk of hemorrhagic transformation and/or poor medical status.
Period: Overall Study
Arm/Group | Conventional | Surgery
Started | 39 | 37
Completed | 39 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional | Surgery | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (17) | 46 (15) | 47 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 27 | 24 | 51
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With In-hospital Death or Clinical Embolic Events
Description: The composite of in-hospital death and clinical embolic events confirmed by imaging studies: the acute onset of clinical symptoms or signs of embolism and the occurrences of new lesions, as confirmed by follow-up imaging studies.
Time Frame: within 6 weeks from the randomization
Population: intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Conventional | Surgery
Number analyzed (Participants) | 39 | 37
participants | 9 | 1
Statistical Analysis 1: Comparison: Conventional vs Surgery; We estimated that a sample size of 74 patients would provide 80% power to detect a significant difference with respect to the primary end point at the 2-sided significance level of 0.05, assuming that the in-hospital event rate would be 23% in the conventional treatment group and 3% in the early surgery group; Test type: Superiority or Other; p < 0.05, Fisher Exact; Hazard Ratio (HR) = 0.10

2. Secondary Outcome: All-cause Death
Time Frame: up to 6 month after enrollment
Reporting Status: Not Posted

3. Secondary Outcome: Recurrences of Infective Endocarditis
Time Frame: up to 6 months after enrollment
Reporting Status: Not Posted

4. Secondary Outcome: All Embolic Events Including Symptomatic and Asymptomatic Embolization Documented by Imaging Studies
Time Frame: up to 6 months after enrollment
Reporting Status: Not Posted

5. Secondary Outcome: Readmission Due to Development of Congestive Heart Failure
Time Frame: up to 6 months after enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All patients underwent complete follow-up that began in September 2006 and ended in September 2011.
Arm/Group | Conventional | Surgery
Serious Adverse Events (participants affected / at risk) | 9/39 | 1/37
Other Adverse Events (participants affected / at risk) | 1/39 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional (N=39) | Surgery (N=37)
Cardiac death (Cardiac disorders) | 2 (2) | 0 (0)
embolism (Vascular disorders) | 8 (8) | 0 (0)
In-hospital noncardiac death (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional (N=39) | Surgery (N=37)
recurrence of infective endocarditis (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The EASE trial was a limited study in scope, in that it included patients with severe valvular disease and large vegetations, and excluded those with major stroke, prosthetic valve endocarditis or aortic abscess.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No